CLINICAL TRIAL: NCT04996290
Title: Combined Pericapsular Nerve Group (PENG) and Lateral Femoral Cutaneous Nerve (LFCN) Block for Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Combined PENG and LFCN Block for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Lennert De Schrijver, Principal Investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3002020000032
Record Dates: First submitted 2021-07-19; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia, Conduction; Pain, Postoperative; Arthroplasty, Replacement, Hip
Keywords: regional anesthesia; postoperative pain; total hip arthroplasty; pericapsular nerve group block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG + LFCN block (Active Comparator): The participants in this group received a combined regional technique just before surgery:
  * Pericapsular nerve group (PENG) block
  * Lateral femoral cutaneus nerve (LFCN) block
  Interventions: Procedure: PENG + LFCN block; Drug: Ropivacaine injection
- No regional anesthesia (No Intervention): Control group

INTERVENTIONS:
Procedure: PENG + LFCN block — Regional anesthesia technique
  Other Names: pericapsular nerve group block; lateral femoral cutaneous nerve block
  Arms: PENG + LFCN block
Drug: Ropivacaine injection — Local anesthetic used for peripheral nerve block.
  Other Names: ropivacaine 0.375%
  Arms: PENG + LFCN block

SUMMARY:
A clinical trial investigating the effect of a combined locoregional anesthesia technique on the postoperative analgesia outcomes after a total hip arthroplasty. A PENG block will be used in combination with a LFCN block. The results will be compared to a control group that is solely treated with intravenous analgesia. This technique aims to provide improved pain scores after surgery without interference of revalidation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who underwent a primary total hip replacement under general anesthesia

Exclusion Criteria:

* insulin dependent diabetes mellitus
* chronic pain
* severe dementia or mental retardation
* allergy to local anesthetics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Initial pain score | 0 hours postoperative
  numeric rating score (NRS) of 0 to 10
Pain score after 2h | 2 hours postoperative
  numeric rating score (NRS) of 0 to 10
Pain score after 24h | 24 hours postoperative
  numeric rating score (NRS) of 0 to 10

SECONDARY OUTCOMES:
Initial motor function | 0 hours postoperative
  score chart inspired by the Bromage score (NRS) of 0 to 3
Motor function after 2h | 2 hours postoperative
  score chart inspired by the Bromage score (NRS) of 0 to 3
Motor function after 24h | 24 hours postoperative
  score chart inspired by the Bromage score (NRS) of 0 to 3
Intraoperative opioids | intraoperative
  dose of intravenous opioids in microgram per kilogram bodyweight
Postoperative opioids | 24 hours postoperative
  dose of intravenous opioids in microgram per kilogram bodyweight

CONTACTS AND LOCATIONS:
Overall Officials: Yzabel Vandevivere, MD, Principal Investigator — AZ Monica
Locations (1):
- AZ Monica, Deurne, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Morrison C, Brown B, Lin DY, Jaarsma R, Kroon H. Analgesia and anesthesia using the pericapsular nerve group block in hip surgery and hip fracture: a scoping review. Reg Anesth Pain Med. 2021 Feb;46(2):169-175. doi: 10.1136/rapm-2020-101826. Epub 2020 Oct 27. PMID 33109730
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Roy R, Agarwal G, Pradhan C, Kuanar D. Total postoperative analgesia for hip surgeries, PENG block with LFCN block. Reg Anesth Pain Med. 2019 Mar 28:rapm-2019-100454. doi: 10.1136/rapm-2019-100454. Online ahead of print. No abstract available. PMID 30923252
- [Background] Hojer Karlsen AP, Geisler A, Petersen PL, Mathiesen O, Dahl JB. Postoperative pain treatment after total hip arthroplasty: a systematic review. Pain. 2015 Jan;156(1):8-30. doi: 10.1016/j.pain.0000000000000003. PMID 25599296